CLINICAL TRIAL: NCT03879499
Title: The Value of Postoperative CRP Levels to Predict Postoperative Vaginal Cuff Hematoma
Brief Title: Postoperative CRP Levels and Vaginal Cuff Hematoma
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Kadirogulları, Principal investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2017/78
Record Dates: First submitted 2019-03-12; First posted 2019-03-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Postoperative Hematoma
Keywords: cuff hematoma; CRP levels

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
After laparoscopic hysterectomy, authors aimed to determine cuff hematoma and a postoperative CRP value to help predict the other complications.

A total of 136 patients who underwent total laparoscopic hysterectomy (TLH) were evaluated. CRP, White blood cell (WBC) and hemoglobin values (Hb) were measured on the 1st, 2nd and 7th days before and after the operation. Complications, pre-postoperative vaginal length and female sexual function were evaluated. Fourteen patients who developed cuff hematoma during postoperative follow-up were analyzed with the receiver operating characteristics (ROC) curve. ROC curves with the largest area under the curve for each inflammatory marker were compared in order to define the marker with higher diagnostic accuracy.

ELIGIBILITY:
Inclusion Criteria:women who underwent TLH operation with benign gynecological indications

Exclusion Criteria:

* Decided to switch to laparotomy during operation
* postoperative complication due to relaparotomy
* infection (including urinary system and lung infections)
* Blood transfusion after TLH
* with rheumatic diseases
* length of hospital stay due to wound infection

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women who underwent TLH operation with benign gynecological indications
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Relationship between CRP Levels and cuff hematoma; crp levels | 1 week
  The value of Postoperative CRP Levels to predict Postoperative Vaginal Cuff Hematoma ; To evaluate tissue trauma and surgical inflammatory responses, venous peripheral blood samples (C-reactive protein) were taken on the first, second and seventh day postoperatively. CRP values were measured under standardized conditions using turbidometry. CRP levels (mg / dl) were recorded.
Relationship between CRP Levels and cuff hematoma; cuff hematoma measurement | 15 days
  The patients were called to the outpatient clinic after the hysterectomy and evaluated by transvaginal ultrasonography (tvusg) for cuff hematoma.hematoma dimensions recorded in centimeters.